CLINICAL TRIAL: NCT05179889
Title: mFOLFIRINOX Versus mFOLFOX 6 as Adjuvant Treatment for High Risk Stage III (pT4N1/2 or pTanyN2) Colon Cancer: Multicenter, Open Labeled, Randomized, Phase II Study
Brief Title: Adjuvant mFOLFIRINOX for High-risk Stage III Colon Cancer
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chungnam National University Hospital (Other)
Collaborators: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Principal Investigator, Kyung-ha Lee, Associate professor, Chungnam National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-11-062
Record Dates: First submitted 2021-12-17; First posted 2022-01-06 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Colon Cancer Stage III
Keywords: High risk stage III (pT4N1/2 or pTanyN2) colon cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): mFOLFIRINOX
  Interventions: Drug: mFOLFIRINOX
- Arm B (Active Comparator): mFOLFOX 6
  Interventions: Drug: mFOLFOX 6

INTERVENTIONS:
Drug: mFOLFIRINOX — Irinotecan 150 mg/m2 IV day 1, oxaliplatin 85 mg/m2 IV day 1, Leucovorin 400 (or levoleucovorin 200) mg/m2 IV day 1, 5-FU 1200 mg/m2/d IV x 2 days (total 2400 mg/m2 over 48 hours) continuous infusion] 12 cycles per 2 weeks
  mFOLFOX 6 [Oxaliplatin 85 mg/m2 IV day 1, Leucovorin 400 (or levoleucovorin 200) mg/m2 IV day 1, 5-FU 400 mg/m2 IV bolus day 1, 5-FU 1200 mg/m2/d IV x 2 days (total 2400 mg/m2 over 46-48 hours) continuous infusion, 12 cycles per 2 week
  Arms: Arm A
Drug: mFOLFOX 6 — Oxaliplatin 85 mg/m2 IV day 1, Leucovorin 400 (or levoleucovorin 200) mg/m2 IV day 1, 5-FU 400 mg/m2 IV bolus day 1, 5-FU 1200 mg/m2/d IV x 2 days (total 2400 mg/m2 over 46-48 hours) continuous infusion, 12 cycles per 2 weeks
  Arms: Arm B

SUMMARY:
A multicenter, open labeled randomized, phase II trial comparing mFOLFIRINOX and mFOLFOX6 as adjuvant treatment for high risk stage III (pT4N1/2 or pTanyN2) colon cancer

DETAILED DESCRIPTION:
After inclusion and exclusion criteria have been fulfilled and the patient consent has been obtained, the patient will be included and randomized to mFOLFIRINOX or mFOLFOX 6 with a 1:1 ratio.

Arm A: mFOLFIRINOX Arm B: mFOLFOX

ELIGIBILITY:
Inclusion Criteria:

1. Age of 20-70 years with an ECOG ≤ 2
2. Age of 71-75 years with an ECOG = 0
3. Pathologically confirmed high-risk stage III colon adenocarcinoma (pT4N1 or pTanyN2)
4. Curative radical resection (successful R0 resection) within 60 days before randomization
5. Adequate organ functions

   * ANC ≥ 2×106 cells/mL
   * Hemoglobin ≥ 9.0 g/dL
   * Platelets ≥ 100×106 cells/mL
   * Alanine aminotransferase/aspartate aminotransferase ≤2.5 × times the upper limit of normal (ULN)
   * Serum total bilirubin ≤ 1.5 ULN
   * Alkaline phosphatase ≤ 2.5 × ULN
   * Serum creatinine ≤1.5 × ULN or creatinine clearance > 50 mL/min (Cockcroft-Gault formula)
6. Able to understand and willing to sign and date written voluntary informed consent form
7. Life expectancy ≥ 5 years

Exclusion Criteria:

1. Distant metastasis
2. Middle or lower rectal cancer of need for radiotherapy
3. Postoperative complication of 3 or more grades of Clavien-Dindo classification
4. Underlying disease or postoperative condition which is contraindication for chemotherapy
5. Known hypersensitivity reaction to any study treatment component
6. Familial adenomatosis polyposis or hereditary non-polyposis colorectal cancer
7. Inflammatory bowel disease
8. Previous other malignancy which cannot be curatively treated
9. Pregnancy or breast feeding
10. Any other situation would exclude the patient from study based on the investigator's opinion

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2021-07-06 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | 3 years after the operation
  the time from the date of operation to the date of the first recurrence or the death from any cause

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years after the operation
  the time from the date of operation to the date of the death from any cause
Incidence of treatment-related adverse events | 3 years after the operation
  Toxicity of all grade and more than grade 3 based on CTCAE version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Ha Lee, Principal Investigator — Chungnam National University Hospital
Locations (1):
- Chungnam National University Hospital, Daejeon, South Korea

REFERENCES:
- [Derived] Lee KH, Yang IJ, Ha GW, Lee J, Park YY, Lee SH, Lee JM, Bae JH, Park EJ, Kim H, Kim KY, An S, Kim IY, Kim JY. mFOLFIRINOX versus mFOLFOX 6 as adjuvant treatment for high-risk stage III colon cancer - the FROST trial: study protocol for a multicenter, randomized controlled, phase II trial. BMC Cancer. 2024 Mar 29;24(1):397. doi: 10.1186/s12885-024-11939-x. PMID 38553680